CLINICAL TRIAL: NCT04225312
Title: Personalized Extended Interval Dosing of Natalizumab in Relapsing Remitting Multiple Sclerosis
Acronym: SUPERNEXT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Stichting MS Research (Unknown); Innovatiefonds Zorgverzekeraars (Other); Stichting Treatmeds (Unknown)
Responsible Party: Principal Investigator, Zoé van Kempen, Principal investigator, Amsterdam UMC, location VUmc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL70503.029.19
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Natalizumab; Extended interval dosing
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Intervention Model Description: Prospective national phase IV natalizumab cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Personalized extended interval dosing (Experimental): Patients will be receiving a personalized dosing schedule from 6 weeks, which will be further extended if the trough level exceeds 10 ug/ml.
  Interventions: Drug: Personalized extended interval dosing of natalizumab
- Standard interval dosing (Other): Patients who prefer to stay on standard interval dosing.
  Interventions: Drug: Standard interval dosing
- Historic cohort (Other): Historic cohort of natalizumab treated patients on standard interval dosing.
  Interventions: Drug: Standard interval dosing

INTERVENTIONS:
Drug: Personalized extended interval dosing of natalizumab — Personalized extended interval dosing of natalizumab with a schedule from every 6 weeks, which will be further extended if the trough level exceeds 10 ug/ml.
  Other Names: EID
  Arms: Personalized extended interval dosing
Drug: Standard interval dosing — Standard interval dosing in control group and historic group
  Other Names: SID
  Arms: Historic cohort; Standard interval dosing

SUMMARY:
Rationale: Natalizumab is an effective drug in the treatment for relapsing remitting multiple sclerosis (RRMS) and is approved by de FDA/EMA in a treatment regimen of 4-weekly 300mg natalizumab infusions. Natalizumab trough concentrations after a 4-weekly interval are high in the large majority of patients which implies a relative overdose in most patients. A recent randomized controlled trial (RCT) suggests natalizumab maintains a high level of effi-cacy in stable patients with RRMS switching to a 6 week interval. Our study group demon-strated that efficacy of natalizumab is maintained when the infusion interval is extended based on natalizumab trough concentrations (personalized extended interval dosing). This leads to fewer hospital visits, a decrease of healthcare costs and decrease of risk of compli-cations of natalizumab treatment.

Objective: Our objective is to test feasibility and validate safety of personalized extended interval dosing of natalizumab starting from 6 weeks in a large real-life cohort across the Netherlands.

Study design: Prospective national phase IV natalizumab cohort study.

Study population: All patients, aged 18 years or older, who are currently treated with natalizumab in the Netherlands for RRMS, with a minimum of 6 consecutive infusions.

Intervention: All patients currently included in the NEXT-MS trial will receive an adjusted personalized extended interval dosing treatment regimen of natalizumab based on natalizumab concentrations starting from an infusion interval of 6 weeks.

Main study parameters/endpoints: Our main study endpoint is the safety (defined by radiological disease activity) of personalized natalizumab dosing in a large real-life cohort across the Netherlands. Data will be collected regarding disease activity and disability progression. A cost analysis will be performed to show the extent of cost reduction. Patients will be annually followed to assess the influence of personalized dosing on JC virus conversion, JC virus index, incidence of progressive multifocal leukoencephalopathy, treatment satisfaction and quality of life. The influence of personalized dosing on pharmacokinetics will be monitored.

DETAILED DESCRIPTION:
This a national open label phase IV natalizumab cohort study. Our aim is that the large majority of natalizumab treated RRMS patients who are currently treated with PEID in The Netherlands will continue in this study with a treatment interval ≥6 weeks. We will continue the NEXT-MS study with 24 participating centers. The study duration is two years. This study will contain the PEID group, a control group and a historic control group. Participants will decide in which group they will participate as this is an open label, non-randomized study. We have chosen this design as we expect the large majority of patients wanting a personalized natalizumab treatment for the following reasons. Others and our own study group have studied personalized and extended dosing of natalizumab treatment, all indicating that this is a safe approach. Data from the NOVA trial support this approach. As we see a drastic reduction of PML risk with extended interval dosing there is a growing trend internationally to personalized/extended interval dosing. Furthermore, there is an increasing wish in patients and physicians for personalized treatment to increase patient convenience and lowering costs of expensive medication and healthcare.

Based on recent data from the NOVA-trial and data from our preliminary analyses, all patients in the PEID group will continue with personalized dosing with an interval ≥6 weeks. The PEID study group will receive a personalized treatment with the aim of a natalizumab trough concentration of 5μg/ml.

If patients do not desire a personalized treatment, they will be asked informed consent for the use of their patient data and for the questionnaires as the control group. As this introduces a bias, the PEID group will be compared to a historical cohort of Amsterdam MS Center.

Furthermore, the patients of the control group will be asked to donate blood once for measuring of natalizumab trough concentration.

As of April 2021, the European Commission has granted marketing authorization for SC in-jection of natalizumab. As pharmacokinetics and pharmacodynamics between SC and IV ad-ministration resulted in comparable trough natalizumab serum concentration and a4-integrin receptor saturation, patients who desire a switch from IV administration to SC administration will have the opportunity to continue the study in the same study group.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remitting multiple sclerosis according to the 2017 criteria
* 6 or more consecutive natalizumab infusions
* 18 years or older
* Agreed to participate (written informed consent)

Exclusion Criteria:

* High titer natalizumab (>100 arbitrary units (AU)/ml) antibodies
* Contraindication for frequent magnetic resonance imaging (MRI) (ie, pacemaker or other contraindicated implanted metal devices, or have claustrophobia that cannot be medically managed)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Change of T2 lesions on brain MRI | Baseline, year 1, year 2
  Assessing new/enlarging T2 lesions on brain MRI

SECONDARY OUTCOMES:
Annualized relapse rate | Baseline, year 1, year 2
  Clinical relapses during personalized extended interval dosing
Disability progression during follow-up | Baseline, year 1, year 2
  Disability progression measured on the Expanded Disability Status Scale (EDSS); running form 0 (no disability) to 10 (death)
Cost analysis | Baseline, year 1, year 2
  Cost-utility analysis using EuroQol 5D (EQ-5D) and the Work Productivity and Activtiy Impairment Questionnaire (WPAI).
JC virus conversion | 6 monthly JCV measurement for two years
  Annual conversion rate of the John Cunningham Virus (JCV)
Course JC virus index | 6 monthly JCV measurement for two years
  Course of John Cunningham Virus (JCV) index in JCV positive patients
Natalizumab wearing-off effect | Baseline, year 1, year 2
  Occurrence of the natalizumab wearing-off effect
Stability of natalizumab trough concentration | 6 monthly natalizumab trough concentrations for two years
  Long-term stability of natalizumab trough concentration in personalized interval dosing
Patient preference | Baseline
  Percentage of patients preferring personalized treatment over standard treatment and percentage staying on personalized treatment
Quality of life: MSIS-29 | Baseline, year 1, year 2
  Quality of life on the Multiple Sclerosis Impact Scale (MSIS-29)
Satisfaction of treatment: TSQM | Baseline, year 1, year 2
  Satisfaction of treatment on the Treatment Satisfaction Questionnaire of Medication (TSQM)
Progressive multifocal leukoencephalopathy | Trough study completion, an average of 2 years
  Incidence of progressive multifocal leukoencephalopathy
Brain atrophy | Baseline, year 1, year 2
  Percentage of patients preferring personalized treatment over standard treatment and percentage staying on personalized treatment
Serum neurofilament light levels | Trough study completion, an average of 2 years
  Difference in serum neurofilament light levels with personalized interval dosing

CONTACTS AND LOCATIONS:
Locations (24):
- Netherlands (24):
  - Jeroen Bosch Hospital, 's-Hertogenbosch
  - Ziekenhuisgroep Twente hospital, Almelo
  - Flevoziekenhuis, Almere Stad
  - Amsterdam UMC, location VUmc, Amsterdam
  - OLVG, Amsterdam
  - Rijnstate Hospital, Arnhem
  - Wilhelmina hospital Assen, Assen
  - Amphia Hospital, Breda
  - Reinier de Graaf hospital, Delft
  - Slingeland Hospital, Doetinchem
  - Ommelander Hospital Groningen, Groningen
  - University Medical Center Groningen, Groningen
  - Spaarne gasthuis hospital, Haarlem
  - Sint-Jansdal Hospital, Harderwijk
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Alrijne Hospital, Leiden
  - Maasstad hospital, Maastricht
  - Canisius Wilhelmina Hospital, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - Haaglanden Medical Center, The Hague
  - Elizabeth tweesteden Hospital, Tilburg
  - Diakonessenhuis, Utrecht
  - St. Antonius Hospital, Utrecht
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foley JF, Defer G, Ryerson LZ, Cohen JA, Arnold DL, Butzkueven H, Cutter G, Giovannoni G, Killestein J, Wiendl H, Smirnakis K, Xiao S, Kong G, Kuhelj R, Campbell N; NOVA study investigators. Comparison of switching to 6-week dosing of natalizumab versus continuing with 4-week dosing in patients with relapsing-remitting multiple sclerosis (NOVA): a randomised, controlled, open-label, phase 3b trial. Lancet Neurol. 2022 Jul;21(7):608-619. doi: 10.1016/S1474-4422(22)00143-0. Epub 2022 Apr 25. PMID 35483387
- [Derived] Toorop AA, van Lierop ZY, Gelissen LM, Hoitsma E, Zeinstra EM, van Rooij LC, van Munster CE, Vennegoor A, Mostert JP, Wokke BH, Kalkers NF, Hoogervorst EL, van Eijk JJ, Roosendaal CM, Kragt JJ, Eurelings M, van Genugten J, Nielsen J, Sinnige L, Kloosterziel ME, Arnoldus EP, van Dijk GW, Bouvy WH, Wessels MH, Boonkamp L, Strijbis EM, van Oosten BW, De Jong BA, Lissenberg-Witte BI, Barkhof F, Moraal B, Teunissen CE, Rispens T, Uitdehaag BM, Killestein J, van Kempen ZL. Prospective trial of natalizumab personalised extended interval dosing by therapeutic drug monitoring in relapsing-remitting multiple sclerosis (NEXT-MS). J Neurol Neurosurg Psychiatry. 2024 Apr 12;95(5):392-400. doi: 10.1136/jnnp-2023-332119. PMID 37963723